CLINICAL TRIAL: NCT01442662
Title: Phase II Multicenter Study to Determine the Efficacy of Gemcitabine With Pazopanib as Second Line Treatment in Patients With Metastatic or Relapsed Uterine or Soft Tissue Leiomyosarcomas
Brief Title: Efficacy of Gemcitabine With Pazopanib as Second Line Treatment in Patient With Metastatic or Relapsed Uterine
Acronym: LMS03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARCOME 11/1101; 2011-001308-36 (EudraCT Number)
Record Dates: First submitted 2011-08-10; First posted 2011-09-28 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Leiomyosarcoma
Keywords: Metastatic or relapsed uterine or soft tissue leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma; Neoplasm Metastasis | interventions — pazopanib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pazopanib, gemcitabine (Experimental): pazopanib tablets (200mg) per os, 800mg/day continuously gemcitabine IV, 2 injection per cycle
  Interventions: Drug: pazopanib + gemcitabine

INTERVENTIONS:
Drug: pazopanib + gemcitabine — pazopanib tablets (200mg) per os, 800mg/day continuously gemcitabine IV, 2 injection per cycle

SUMMARY:
The aim of this research is to study the activity of pazopanib in second line after anthracyclines in extra uterus and uterine LMS in association with gemcitabine.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the PFS using combination of gemcitabine and pazopanib in patients with metastasis or relapse leiomyosarcoma (uterine or soft tissue)who have already received s first line anthracycline based therapy.

Secondary objectives:

To determine the disease control rate To determine the response rate To determine toxicities associated with combined gemcitabine and pazopanib To determine correlation between metabolic response and PFS

Design:

All eligible patients entering the study will receive daily oral pazopanib at 800mg, supplied as 200 mg aqueous film-coated tablets and 2 intravenous gemcitabine every three weeks (8 cycles max).

The treatment will continue until the development of unacceptable toxicity or evidence of disease progression or until patient's / investigator's decision of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of metastatic or relapsed of uterine or soft tissue leiomyosarcoma previously treated with one line of chemotherapy with at least an anthracycline. Patients who have received adjuvant therapy less than one year before relapse were considered to have received a first line therapy for metastatic disease)
* Delay between the end of previous treatment (chemotherapy, hormonotherapy, radiotherapy, immunotherapy, surgery or tumor embolisation) must be > 4 weeks
* At least one measurable lesion with RECIST criteria with progressive disease between the last 6 weeks between inclusion. One target at least must be in a non irradiated area
* performance status ECOG ≤ 2
* Age ≥ 18 years
* Subjects must provide written informed consent prior to performance of study-specific procedures, and must be willing to comply with treatment and follow up
* Adequate hematologic function
* Adequate coagulation function
* Adequate renal function
* Adequate liver function
* Patients must be affiliated to a Social Health Insurance
* Women of childbearing potential must be using a medically accepted method of contraception and must have a negative serum pregnancy test within 14 days of enrollment and/or urine pregnancy test 72 hours prior to the administration of the first study treatment.
* LVEF ≥ site limits

Main Exclusion Criteria:

* Other uterine or soft tissue sarcomas
* Symptomatic or known brain metastasis
* Radiation therapy on the only evaluable lesion
* Anti coagulant treatment
* strong inhibitors or inducers of the isoenzyme CYP3A4 treatment
* Known sero-positivity (HIV, HbC, HbS)or uncontrolled infection
* other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* Clinically significant gastrointestinal abnormalities that may affect the absorption of the IP
* Corrected QT interval > 480 msec
* Other serious underlying pathology that would preclude study treatment
* Calcium and magnesium levels inferior to standard levels (measured within 14 days before the first pazopanib dose) and potassium levels inferior to standard levels (measured within 72 hours before the first pazopanib dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 9 months
  To assess the 9-month Progression Free Survival in Patients With Metastatic or Relapsed Uterine or Soft Tissue Leiomyosarcomas and treated with Gemcitabine and Pazopanib

SECONDARY OUTCOMES:
disease control rate and overall response rate | 12 weeks
Safety of the combination Gemcitabine-Pazopanib | during the entire trial
  The severity of the adverse events and toxicity will be graded according to the NCI CTC-AE v4.0
metabolic response by using PET scan | 6 weeks
  First PET scan at baseline and the second one at 6 weeks after the first administration

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pautier, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (17):
- France (17):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre G.F Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Timone, Marseille
  - Centre Val d'Aurelle Paul Lamarque, Montpellier
  - Institut de Cancérologie de l'Ouest/Centre René Gauducheau, Nantes Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Hôpital Claudius Regaud, Paris
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hopital René Huguenin, Saint-Cloud
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
PD will not be shared at an individual level, they will be part of the study database including all enrolled patients

REFERENCES:
- [Derived] Pautier P, Penel N, Ray-Coquard I, Italiano A, Bompas E, Delcambre C, Bay JO, Bertucci F, Delaye J, Chevreau C, Cupissol D, Bozec L, Eymard JC, Saada E, Isambert N, Guillemet C, Rios M, Piperno-Neumann S, Chenuc G, Duffaud F. A phase II of gemcitabine combined with pazopanib followed by pazopanib maintenance, as second-line treatment in patients with advanced leiomyosarcomas: A unicancer French Sarcoma Group study (LMS03 study). Eur J Cancer. 2020 Jan;125:31-37. doi: 10.1016/j.ejca.2019.10.028. Epub 2019 Dec 10. PMID 31835236